CLINICAL TRIAL: NCT02576691
Title: Effects of Percutaneous Coronary Intervention in Patients With Cardiac Arrest After Acute Myocardial Infarction: a 2-Year Study
Status: Completed | Type: Observational
Sponsor: Yuanli Lei (Other)
Responsible Party: Sponsor-Investigator, Yuanli Lei, First Affiliated Hospital of Wenzhou Medical University, Yuanli Lei, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Other Study IDs: Yuanli2015
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Acute Myocardial Infarction
Keywords: cardiac arrest; percutaneous coronary intervention; cardiogenic shock; outcome
MeSH Terms: conditions — Heart Arrest; Shock, Cardiogenic | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- The PCI group: The PCI group was composed of patients who underwent PCI following the return of spontaneous circulation or after CA.
  Interventions: Device: percutaneous coronary intervention
- Non-PCI group: Non-PCI group included patients who didn't undergo PCI or were subjected to PCI before CA

INTERVENTIONS:
Device: percutaneous coronary intervention
  Groups: The PCI group

SUMMARY:
The purpose of this study is To assess percutaneous coronary intervention 's effect on short- and long- term outcomes, and complication incidence in resuscitated victims of cardiac arrest after acute myocardial infarction

ELIGIBILITY:
Inclusion Criteria:

* underwent successful cardiopulmonary resuscitation from CA after AMI

Exclusion Criteria:

* late tumor;
* underwent Coronary Artery Bypass Grafting after CAG;
* with no attempted resuscitation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 20 million residents of the South of Zhejiang Province
Sampling Method: Probability Sample
Enrollment: 2363 (Actual)
Dates: Start 2005-01; Primary Completion 2013-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
all cause mortality | 2 years